CLINICAL TRIAL: NCT00603408
Title: Effect of Neoadjuvant Cisplatin Based Chemoradiation Therapy for Locally Advanced Triple Negative Breast Cancer: Clinical Outcome and Correlation to Biological Parameters
Brief Title: Effect of Chemotherapy and Radiation Prior to Surgery for Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued due to lack of accrual.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0913
Record Dates: First submitted 2007-12-28; First posted 2008-01-29 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Locally Advanced; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Radiotherapy; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin + Radiation + Recommended Surgery (Experimental): Cisplatin 75 mg/m^2 IV Day 1 Week 1, Day 1 Week 2, Day 1 Week 7, Day 1 Week 10
  Radiation = Total dose to breast or chest wall will be 50-60 Gy in 1.8-2.0 Gy daily fractions. Internal mammary nodes, supraclavicular fossa nodes and axillary nodal basins will receive 45-50 Gy over 5-6 weeks.
  Surgery (recommended) mastectomy with/without axillary lymph node dissection
  Interventions: Drug: Cisplatin; Radiation: Radiation Therapy; Procedure: Mastectomy

INTERVENTIONS:
Drug: Cisplatin
  Other Names: cisplatinum
Radiation: Radiation Therapy
Procedure: Mastectomy — (RECOMMENDED BUT NOT REQUIRED)

SUMMARY:
The purpose of this study is to determine whether Cisplatin when given with radiation therapy prior to surgery is effective in improving response to treatment in breast cancer patients. Tumor, blood and bone marrow samples will be collected in this study and will also help researchers determine if cisplatin is able to change tumor DNA so it cannot multiply itself and create more tumor cells, and cause the tumor cells to die.

DETAILED DESCRIPTION:
After Diagnosis: Clinical Stage IIB, III Breast Cancer, Triple Negative

Week 0: Port-A-Cath placement Tumor biopsy (Core and FNA) Blood collection Bone marrow aspiration Sentinel Lymph node biopsy, if axillary US negative

Week 1: Chemo & Radiation Day 1: Radiation Therapy, Cisplatin 75mg/m^2 (cycle 1) Days 2-5: Radiation Therapy

Week 2: Radiation Day 1-5: Radiation Therapy

Week 3: Radiation Days 1-5: Radiation Therapy

Week 4: Chemo & Radiation Day 1: Radiation Therapy, Cisplatin 75mg/m^2 (cycle 2) Days 2-5: Radiation Therapy

Week 5: Radiation Days 1-5: Radiation Therapy

Week 6: Radiation Days 1-5: Radiation Therapy

Week 7: Chemo Day 1: Cisplatin 75mg/m^2 (cycle 3)

Week 10: Chemo Day 1:Cisplatin 75mg/m^2 (cycle 4)

Week 13: Surgery Mastectomy with/without axillary lymph node dissection Tumor biopsy (Core and FNA) Blood collection Bone marrow aspiration

Week 15 - 21: Recommended (physician discretion) Adjuvant Chemo Dose dense Doxorubicin: 60mg/m^2 & Cyclophosphamide: 600mg/m^2, every 2 weeks for 4 cycles

Week 21 - 29: Recommended (physician discretion) Adjuvant Chemo Paclitaxel: 175mg/m^2 every 2 weeks for 4 cycles

Week 52 IVAD Removal, Bone marrow aspiration

Follow-Up (up to 5 years) Q 3 months for year 1 Q 6 months for year 2-3 Q 1 year for years 4-5

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 18 years of age
* Patients must be newly diagnosed with primary invasive ductal breast adenocarcinoma.
* Tumor classified as clinically stage T2, T3 or T4 with any N (NX, N1, N2, or N3).
* Tumor does not express the following biomarkers: estrogen receptor, progesterone receptor, Her2/neu
* Adequate organ function defined as:

  * Serum Creatinine <= 1.5 x upper limit of institutional normal.
  * ALT, AST, ALK Phos <= 1.5 x upper limit of institutional normal.
  * Bilirubin <= 1.5 x upper limit of institutional normal.
  * Normal left ventricular function (LVEF > 50%) by MUGA or ECHO.

Exclusion Criteria:

* No evidence of distant metastasis present by CT, Bone scan, or physical exam. If the bone scan or CT scans demonstrate indeterminate lesions, the nature of these lesions should be further clarified by additional testing such as PET or MRI.
* No prior malignancies with the exception of curatively treated basal or squamous carcinoma of the skin or history of previous malignancies, treated with at least greater than 5 years disease free survival.
* Women of child bearing potential may not be currently pregnant or breastfeeding at time of registration and must agree to use adequate contraception.
* Karnofsky Performance Status of <= 70.
* Patients with known history neural deficiencies (e.g. peripheral neuropathy).
* Patients with a known hearing impairment (hearing loss or severe tinnitus).
* Male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Aft, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Cleator S, Heller W, Coombes RC. Triple-negative breast cancer: therapeutic options. Lancet Oncol. 2007 Mar;8(3):235-44. doi: 10.1016/S1470-2045(07)70074-8. PMID 17329194
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815
- [Background] Carey LA, Perou CM, Livasy CA, Dressler LG, Cowan D, Conway K, Karaca G, Troester MA, Tse CK, Edmiston S, Deming SL, Geradts J, Cheang MC, Nielsen TO, Moorman PG, Earp HS, Millikan RC. Race, breast cancer subtypes, and survival in the Carolina Breast Cancer Study. JAMA. 2006 Jun 7;295(21):2492-502. doi: 10.1001/jama.295.21.2492. PMID 16757721
- [Background] Turner NC, Reis-Filho JS. Basal-like breast cancer and the BRCA1 phenotype. Oncogene. 2006 Sep 25;25(43):5846-53. doi: 10.1038/sj.onc.1209876. PMID 16998499
- [Background] Turner NC, Reis-Filho JS, Russell AM, Springall RJ, Ryder K, Steele D, Savage K, Gillett CE, Schmitt FC, Ashworth A, Tutt AN. BRCA1 dysfunction in sporadic basal-like breast cancer. Oncogene. 2007 Mar 29;26(14):2126-32. doi: 10.1038/sj.onc.1210014. Epub 2006 Oct 2. PMID 17016441
- [Background] Garber, J., Richardson, A., Harris, L., Miron, A., Silver, D., Golshan, M., Ryan, P., Ganesan, S., Wang, Z., Clarke, K., Inglehart, J., and Winer, E. Neoadjuvant cisplatin in triple negative breast cancer. SABCS, 2006.
- [Background] Bollet MA, Sigal-Zafrani B, Gambotti L, Extra JM, Meunier M, Nos C, Dendale R, Campana F, Kirova YM, Dieras V, Fourquet A; Institut Curie Breast Cancer Study Group. Pathological response to preoperative concurrent chemo-radiotherapy for breast cancer: results of a phase II study. Eur J Cancer. 2006 Sep;42(14):2286-95. doi: 10.1016/j.ejca.2006.03.026. Epub 2006 Aug 8. PMID 16893641
- [Background] Formenti SC, Volm M, Skinner KA, Spicer D, Cohen D, Perez E, Bettini AC, Groshen S, Gee C, Florentine B, Press M, Danenberg P, Muggia F. Preoperative twice-weekly paclitaxel with concurrent radiation therapy followed by surgery and postoperative doxorubicin-based chemotherapy in locally advanced breast cancer: a phase I/II trial. J Clin Oncol. 2003 Mar 1;21(5):864-70. doi: 10.1200/JCO.2003.06.132. PMID 12610186
- [Background] Whitney CW, Sause W, Bundy BN, Malfetano JH, Hannigan EV, Fowler WC Jr, Clarke-Pearson DL, Liao SY. Randomized comparison of fluorouracil plus cisplatin versus hydroxyurea as an adjunct to radiation therapy in stage IIB-IVA carcinoma of the cervix with negative para-aortic lymph nodes: a Gynecologic Oncology Group and Southwest Oncology Group study. J Clin Oncol. 1999 May;17(5):1339-48. doi: 10.1200/JCO.1999.17.5.1339. PMID 10334517
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Keys HM, Bundy BN, Stehman FB, Muderspach LI, Chafe WE, Suggs CL 3rd, Walker JL, Gersell D. Cisplatin, radiation, and adjuvant hysterectomy compared with radiation and adjuvant hysterectomy for bulky stage IB cervical carcinoma. N Engl J Med. 1999 Apr 15;340(15):1154-61. doi: 10.1056/NEJM199904153401503. PMID 10202166
- [Background] Rowinsky EK, Donehower RC. Paclitaxel (taxol). N Engl J Med. 1995 Apr 13;332(15):1004-14. doi: 10.1056/NEJM199504133321507. No abstract available. PMID 7885406
- [Background] Rowinsky EK, Chaudhry V, Forastiere AA, Sartorius SE, Ettinger DS, Grochow LB, Lubejko BG, Cornblath DR, Donehower RC. Phase I and pharmacologic study of paclitaxel and cisplatin with granulocyte colony-stimulating factor: neuromuscular toxicity is dose-limiting. J Clin Oncol. 1993 Oct;11(10):2010-20. doi: 10.1200/JCO.1993.11.10.2010. PMID 7692001
- [Background] Diel IJ, Cote RJ. Bone marrow and lymph node assessment for minimal residual disease in patients with breast cancer. Cancer Treat Rev. 2000 Feb;26(1):53-65. doi: 10.1053/ctrv.1999.0150. PMID 10660491
- [Background] Braun S, Pantel K, Muller P, Janni W, Hepp F, Kentenich CR, Gastroph S, Wischnik A, Dimpfl T, Kindermann G, Riethmuller G, Schlimok G. Cytokeratin-positive cells in the bone marrow and survival of patients with stage I, II, or III breast cancer. N Engl J Med. 2000 Feb 24;342(8):525-33. doi: 10.1056/NEJM200002243420801. PMID 10684910
- [Background] Braun S, Naume B. Circulating and disseminated tumor cells. J Clin Oncol. 2005 Mar 10;23(8):1623-6. doi: 10.1200/JCO.2005.10.073. No abstract available. PMID 15755968
- [Background] Janni W, Rack B, Schindlbeck C, Strobl B, Rjosk D, Braun S, Sommer H, Pantel K, Gerber B, Friese K. The persistence of isolated tumor cells in bone marrow from patients with breast carcinoma predicts an increased risk for recurrence. Cancer. 2005 Mar 1;103(5):884-91. doi: 10.1002/cncr.20834. PMID 15666325
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cisplatin + Radiation + Recommended Surgery: Cisplatin 75 mg/m2 IV Day 1 Week 1, Day 1 Week 2, Day 1 Week 7, Day 1 Week 10
  Radiation = Total dose to breast or chest wall will be 50-60 Gy in 1.8-2.0 Gy daily fractions. Internal mammary nodes, supraclavicular fossa nodes and axillary nodal basins will receive 45-50 Gy over 5-6 weeks.
  Surgery (recommended) mastectomy with/without axillary lymph node dissection
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 52 [42 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: * Complete response: disappearance of all target lesions, non-target lesions, and normalization of tumor marker level
  * Partial response: at least a 30% decrease in the sum of the longest diameter (LD) of the target lesions taking as reference the baseline sum LD
  * Stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started,
  * Progressive disease: at least a 20% increase in the sum of the LD of the target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, appearance of one more new lesions, or unequivocal progression of existing non-target lesions.
Time Frame: At the time of surgery (week 13)
Measure: Number; unit: participants
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 5
participants
  Complete response | 2
  Partial response | 3
  Stable disease | 0
  Progressive disease | 0

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression: time from registration until objective tumor progression; does not include deaths
Time Frame: Until study was terminated (23.5 months)
Population: At the time of study termination, no participants had experienced disease progression.
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival Rate (OS)
Description: OS = Time from registration until death from any cause
Time Frame: Until study was terminated (23.5 months)
Measure: Number; unit: percentage of participants
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 5
percentage of participants | 100

4. Secondary Outcome: Number of Participants With Surgical Complications
Time Frame: 30 days post surgery (week 17-18)
Measure: Number; unit: participants
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 5
participants | 0

5. Secondary Outcome: Number of Participants With Medical Toxicities
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for all toxicity reporting. All detailed information regarding serious and other adverse events are listed in the Adverse Event module of these results.
Time Frame: 30 days post surgery (week 17-18)
Measure: Number; unit: participants
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 5
participants | 5

6. Secondary Outcome: Effect of Neoadjuvant Chemoradiation Therapy in Disseminated Cancer Cells in the Bone Marrow and Correlation to Tumor Response
Time Frame: 5 years
Population: Collecting bone marrow samples were optional and at the time of surgery only 2 patients participated and at the time of port removal submission none of the patients participated.
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 0

7. Secondary Outcome: Develop Animal Models of Triple Negative Breast Cancers
Time Frame: 5 years
Population: Collecting tissue from the optional mastectomy was optional and was not collected on any of the patients.
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 0

8. Secondary Outcome: Provide Samples for the Development of the FNA Assay
Time Frame: At time of IVAD placement and at time of surgery
Population: Collecting tissue from the optional mastectomy was optional and was not collected on any of the patients.
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cisplatin + Radiation + Recommended Surgery
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Radiation + Recommended Surgery (N=5)
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Viral hepatitis (Infections and infestations) | 1
Infection unknown ANC - general wound (Infections and infestations) | 1
Burn due to radiation therapy (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Radiation + Recommended Surgery (N=5)
Allergic reaction (Immune system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (Investigations) | 2
Lymphopenia (Investigations) | 4
Neutrophils (Investigations) | 1
Platelets (Investigations) | 2
Cardiac General - Other (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
INR (Investigations) | 1
PTT (Investigations) | 2
Constitutional symptoms - other (General disorders) | 1
Fatigue (General disorders) | 5
Insomnia (Psychiatric disorders) | 1
Rigors/chills (General disorders) | 1
Alopecia (Social circumstances) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Dermatology - other (Skin and subcutaneous tissue disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation therapy (Skin and subcutaneous tissue disorders) | 5
Hot flashes (Vascular disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Hemmorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Taste alteration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Hematoma (Vascular disorders) | 1
Edema: head and neck (General disorders) | 1
Edema: limb (General disorders) | 3
Lymphatics - other (specify) (Blood and lymphatic system disorders) | 1
Albumin, serum-low (Metabolism and nutrition disorders) | 2
Alkaline phosphatase (Investigations) | 3
ALT (Investigations) | 3
AST (Investigations) | 1
Bilirubin (Investigations) | 1
Creatinine (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Investigations) | 3
Extremity - upper (function) (Musculoskeletal and connective tissue disorders) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mood alteration - anxiety (Psychiatric disorders) | 2
Mood alteration - depression (Psychiatric disorders) | 1
Neuropathy - sensory (Nervous system disorders) | 1
Ocular - other (specify) (Eye disorders) | 1
Pain - general (Pain NOS) (General disorders) | 1
Pain - General (tumor pain) (General disorders) | 1
Pain - musculoskeletal (joint) (Musculoskeletal and connective tissue disorders) | 2
Pain - musculoskeletal (neck) (Musculoskeletal and connective tissue disorders) | 1
Pain - Neurology (head/headache) (Nervous system disorders) | 1
Pain - Other (specify) (General disorders) | 2
Pain - Pulmonary (chest wall) (Respiratory, thoracic and mediastinal disorders) | 1
Pain - Pulmonary (Chest/thorax NOS) (Respiratory, thoracic and mediastinal disorders) | 2
Pain - Sexual (breast) (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Sexual - Other (specify) (Reproductive system and breast disorders) | 1
Vaginitis (Reproductive system and breast disorders) | 1
Surgery Injury - skin (breast) (Injury, poisoning and procedural complications) | 1
Phlebitis (Vascular disorders) | 1
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes